CLINICAL TRIAL: NCT05099679
Title: A Pilot Study for Optimizing Mental Wellbeing and Heart Health for Black Patients With Prostate Cancer
Brief Title: Pilot Study for Black Men With Prostate Cancer: Optimization Of Mental and Heart Health, the BOOM-Heart Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alice Fan, Associate Professor of Medicine (Oncology) and, by courtesy, of Urology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-60375; PROS0109 (Other: Stanford); NCI-2022-02832 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-10-11; First posted 2021-10-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial intervention + Cardiac Rehab Services (Other): Cognitive Behavioral Therapy + Cardiac Rehab
  Interventions: Behavioral: Cognitive behavioral therapy (supportive counseling); Behavioral: Virtual Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (supportive counseling) — Patients will complete a psychosocial intake that generally takes up to 2 hours, but the time required for the intake varies per patient. Subsequently they will be offered up to 7 optional counseling sessions with a clinical social worker
Behavioral: Virtual Cardiac Rehabilitation — If eligible, patients will be referred to Movn Health Virtual Cardiac Rehabilitation to provide approximately 3 exercise sessions per week, with approximately eight coaching sessions over a 12 week period

SUMMARY:
Pilot study to determine the feasibility of providing psychosocial and cardiac rehabilitation services to address socioeconomic health disparities and improve wellbeing for black men with prostate cancer.

DETAILED DESCRIPTION:
Subjects will see an oncology Associate Clinical Social Worker at Stanford's Cancer Center for a two hour psychosocial assessment. Subsequently participants will complete the psychosocial intake support session and elective additional counseling sessions (Part A) at the end of up to 8 counseling sessions (maximum sessions possible) or 20 weeks (+/- 4 weeks), whichever comes first. For participants who continue onto cardiac services (Part B), the participant will complete the cardiac rehabilitation exercise program within 12 weeks (+/- 2 weeks) of the first day of exercise start. The end of study will occur after the last cardiac rehabilitation exercise session (+ 2 weeks).

ELIGIBILITY:
Inclusion Criteria for Part A (Mental Health Services)

* Self-Identify as Black and/or African American.
* Diagnosed with prostate cancer currently or any time in the past (per medical history; pathology not required, active prostate cancer at time of enrollment is not required).
* Males >= age 18.
* All participants must have a life expectancy of > 6 months.
* Participants must have the ability to understand and the willingness to sign a written informed consent document in English, and the willingness/ability to comply with the protocol activities.
* Ability to wear a face mask during all in-person sessions (when required).

Participants must complete the psychosocial intake (Part A, Visit A1) in order to enroll in a cardiac rehabilitation program (Part B).

Additional Inclusion Criteria for Part B (Cardiac Services)

* Have completed the psychosocial intake portion of Visit A1 (as documented by clinical social worker).
* Meets at least one of the following ([a] or [b]):

  1. planning to receive androgen deprivation on Day 1, or is currently, or was formerly, on androgen deprivation therapy. It is acceptable for participant to switch/transition to another form of androgen deprivation therapy while in the study. Participant may be receiving or planning to receive additional systemic therapy concurrent with androgen deprivation.

     ^ treatment with single agent testosterone-blocking agents (such as, but not limited to bicalutamide) will also be eligible

     OR
  2. patients with a cardiac risk factor may enroll. Cardiac risk factors include, but are not restricted to: pre-hypertension, hypertension, metabolic syndrome, tobacco history, coronary artery disease, CVA/TIA, peripheral vascular disease, obesity, hypercholesterolemia, hyperglycemia, heart failure, or any other cardiac condition based on the discretion of the investigators.
* Participants must have an ECOG Performance Status of <= 2 or at the investigator's discretion, will have the ability to participate in a cardiac rehab program.
* Participants must be able and willing to follow the cardiac rehabilitation activities.
* Participant must have a smartphone or tablet to use for the cardiac rehabilitation app.

Exclusion Criterion for Part A (Mental Health Services)

* Actively engaging in self harm, or currently on a 5150 or 5250.

Exclusion Criteria for Part B (Cardiac Services)

* Uncontrolled angina, active acute coronary syndrome (e.g., unstable angina or acute MI) or poorly controlled arrhythmias.
* In the opinion of the Principal Investigator, have a clinically significant comorbid disease that is likely to affect the ability of the patient to complete the trial, interfere with their ability with measurement of self-reported outcomes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-Identify as Black and/or African American
Enrollment: 14 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of Completers | 12 weeks
  Proportion of screened eligible participants who complete the initial 2-hour psychosocial support session intake.
  The pilot study is considered feasible if the primary endpoint is met in at least 50% of patients. We will evaluate the 95% CI of the feasibility rate.

SECONDARY OUTCOMES:
Difference in Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
Difference of General Anxiety Disorder-7 (GAD-7) score | 12 weeks
Difference of Functional Assessment of Cancer Therapy-Prostate (FACT-P) score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice C Fan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No